CLINICAL TRIAL: NCT06807164
Title: Serratus Plane Block (SPB) Versus Capsaïcine Versus Botox-A for Chronic Neuropathic Pain in Post-mastectomy Syndrome
Acronym: SerCaBot
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Ligue contre le cancer, France (Other); Santelys Association (Other); CTD-CNO, Caen (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SerCaBot-2302
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Post-Mastectomy Neuropathic Pain Syndrome
Keywords: Breast cancer; Chronic neuropathic pain; Post-mastectomy pain; Serratus Plane Block (SPB); Capsaicin; Pain management; Botulinum toxin type A
MeSH Terms: conditions — Breast Neoplasms; Agnosia | interventions — Capsaicin; Transdermal Patch; Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: Phase 2, randomized clinical trial, open-label, evaluating 3 interventions : Capsaicin, Botox-A, SPB
Masking Description: N/A (since the study is open label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Capsaicin 8% Patch (Control) (Active Comparator): Participants in this arm will receive an 8% capsaicin patch in a single treatment session in addition to a systemic treatment that has been ongoing for at least 4 weeks. If pain persists, the capsaicin patch application may be repeated at 12 weeks.
  Interventions: Drug: Capsaicin 8% Patch
- Serratus Plane Block (SPB) (Experimental): Participants in this arm will undergo a Serratus Plane Block (SPB), a local anesthetic injection administered by a trained anesthesiologist, in addition to a systemic treatment that has been ongoing for at least 4 weeks. The SPB can be repeated every two weeks up to a maximum of four sessions within the initial 8-week period if pain persists. A repeat treatment may be considered at 12 weeks if further pain control is needed. This intervention aims to provide extended pain relief for neuropathic pain in post-mastectomy patients
  Interventions: Procedure: Serratus Plane Block
- Botulinum Toxin A (Botox-A) Injection (Experimental): This arm involves administration of Botulinum Toxin A (Botox-A) at the site of pain, in addition to a systemic treatment that has been ongoing for at least 4 weeks. If pain remains unresolved, the injection may be repeated at 12 weeks. Botox-A is used here as a local, long-lasting analgesic intervention aimed at reducing chronic neuropathic pain in patients post-mastectomy.
  Interventions: Procedure: Botulinum Toxin A

INTERVENTIONS:
Drug: Capsaicin 8% Patch — One or two capsaicin patch (8%) are applied for 60 minutes to the site of neuropathic pain, in day-hospital. An oral, antalgic pre-medication may be done with one of the following medications (alone or association): paracetamol 1g, nefopam 30 mg, tramadol 100 mg, morphine 10mg, oxycodone 5mg. Capsaicin will be administered in addition to a systemic treatment that has been ongoing for at least 4 weeks. If pain persists, the capsaicin patch application may be repeated at 12 weeks.
  Other Names: Qutenza®
  Arms: Capsaicin 8% Patch (Control)
Procedure: Serratus Plane Block — The Serratus Plane Block (SPB) is a nerve block performed by a trained anesthesiologist to provide localized pain relief. It involves the injection of a local anesthetic: Maximum 150 mg naropeine combined with 150 μg clonidine hydrochloride into the serratus anterior plane under ultrasound guidance. An anesthesiologist will perform the procedure in a post-interventional recovery room, with light sedation.The SBP will be carried out in addition to a systemic treatment that has been ongoing for at least 4 weeks. The SPB may be repeated every two weeks up to four times in the initial 8-week period, with an additional repeat at 12 weeks if pain control remains insufficient.
  Other Names: SPB
  Arms: Serratus Plane Block (SPB)
Procedure: Botulinum Toxin A — Botulinum Toxin A (Botox-A) is injected into the affected area, with a total of 300 units administered across up to 60 injection sites. An anesthesiologist will perform the procedure in a post-interventional recovery room, with light sedation. This intervention will be carried out in addition to a systemic treatment that has been ongoing for at least 4 weeks, and is aimed at providing prolonged pain relief for post-mastectomy neuropathic pain. Light sedation is provided, and injections may be repeated at 12 weeks if necessary.
  Other Names: Botox-A; Botox
  Arms: Botulinum Toxin A (Botox-A) Injection

SUMMARY:
The goal of this phase II clinical trial is to study the effectiveness of a treatment with Serratus Plane Block (SPB) or Botox-A in comparison with capsaicin for the control of chronic neuropathic pain of post-mastectomy syndrom, that is not adequately managed by systemic treatment alone. The primary outcome will be the pain evaluation at 8 weeks.

123 patients with chronic neuropathic pain of post-mastectomy syndrom insufficiently relieved by systemic treatment alone will be recruited over 24 months at the Centre Oscar Lambret.

Patients will be randomly assigned to one of three treatment groups (41 patients per group):

Capsaicin Botulinum toxin A SPB

Patients will be followed for 24 weeks after the study treatment. The follow-up will include remote evaluation and 2 medical visits during which pain and quality of life will be assessed.

DETAILED DESCRIPTION:
SerCaBot is a randomized, open-label, phase II clinical trial designed to evaluate the efficacy of a treatment with Serratus Plane Block (SPB) or Botox-A compared to capsaicin for the control of chronic neuropathic pain of post-mastectomy syndrom, that is not adequately managed by systemic treatment alone.

123 patients with will be recruited over 24 months at the Centre Oscar Lambret.

This clinical trial will be proposed to patients with chronic neuropathic pain of post-mastectomy syndrome that is not adequately managed by systemic treatment alone.

After consent, an inclusion assessment will be carried out including clinical examination, anamnesis, pain assessment (questionnaires PCS, NPS, DN4, NPSI and collect of antalgic treatment) and evaluation of quality of life (questionnaire SF12) and depression (questionnaire HADS).

Patients will then be randomly assigned to one of three treatment groups : Capsaicin, Botox-A, SPB (41 patients per group). The randomization will be balanced 1:1:1, controlled by minimisation (with a random factor set at 0.8) for the distribution of the following factors:

* Pain level at enrolment (continuous NPS)
* Axillary dissection (yes vs. no)
* Loco-regional adjuvant radiotherapy (yes vs. no)
* Prior change of systemic treatment (yes vs. no)

The study treatment will be administered 1 to 2 weeks after randomization. Treatment will be stopped prematurely in the event of unacceptable toxicity or complication. In each group, a repeat of the treatment may be considered after 12 weeks if further pain control is required. In the SPB group, a repeat is also possible every 2 weeks.

Patients will be followed for 24 weeks after the study treatment. Follow-up will include:

* 2 medical visits at 8 weeks and at 24 weeks including pain assessment (questionnaires NPS, NPSI, record of antalgic treatment), record of adverse events related to study treatment and assessment of quality of life (SF12 questionnaire) and depression (questionnaire HADS).
* remote assessment at week-1, week-2, week-4 and week-6 including assessment of pain (questionnaires NPS, NPSI, record of antalgic treatment) and record of adverse events. This remote assessment will be repeated in case of repetition of treatment at week 12.

Patients will withdraw from the study after the 24 week medical visit. Early withdrawal will be possible in case of patient's decision of withdrawal, breast surgery during follow-up, or death.

ELIGIBILITY:
Inclusion Criteria :

1. Women aged ≥ 18 years;
2. Unilateral breast cancer treated by total or partial mastectomy:

   * with sentinel lymph node technique (SLN) or axillary dissection;
   * with or without immediate reconstruction using a prosthesis;
   * associated or not with radiotherapy and/or chemotherapy;
3. Presenting moderate to severe chronic neuropathic pain, defined by:

   * Numerical Pain Scale (NPS) ≥ 3 and DN4 ≥ 4,
   * on a localised aera ((≤ 240 cm²), at the surgical site, in the axillary hollow, or on the inner side of the ipsilateral arm,
   * between 3 and 9 months after breast surgery,
   * with indication of additional locoregional treatment in complement to a systemic treatment of chronic neuropathic pain, as recommended by the SFETD - French Society for the Study and Treatment of Pain (tricyclic antidepressants or IRSNA or gabapentinoid PLUS lidocaine patch, at the appropriate dosage) and implemented for at least 4 weeks;
4. Patient affiliated with a health insurance plan;
5. Patient informed and having consented to participate in the trial.

Exclusion Criteria :

1. Ipsilateral breast cancer recurrence, regardless of the first treatment;
2. History of breast or thoracic surgery prior to mastectomy with residual pain;
3. Painful polyneuropathy related to chemotherapy requiring treatment;
4. Ongoing or planned loco-regional adjuvant radiotherapy within the next 8 weeks;
5. Treatment area not suitable for potential botulinum toxin type A treatment;
6. Breast reconstruction using flap or lipomodelling;
7. Indication for breast reconstruction within the next 8 weeks;
8. Chronic pain of another etiology such as:

   * Neuropathic pain secondary to a neuroma (localized pain),
   * Radiodermatitis,
   * Phantom breast pain,
   * Lymphedema,
   * Complex regional pain syndrome,
   * Adhesive capsulitis,
   * Fibromyalgia;
9. Hypersensitivity or allergy to anesthetics, capsaicin, naropein, clonidine hydrochloride, an amide-type local anesthetic, botulinum toxin type A, or any excipient contained in the preparations;
10. Infection or inflammation at the injection site;
11. Therapeutic/effective anticoagulation;
12. Clinical signs or medical history leading to the diagnosis of:

    * Hemostasis disorder,
    * Local infection,
    * Severe renal insufficiency (creatinine clearance < 30 mL/min),
    * Thrombocytopenia < 50,000 platelets/mm3;
13. Generalized muscle activity disorders (e.g., myasthenia, Lambert-Eaton syndrome);
14. Heart rate lower than 60/minute;
15. Severe bradyarrhythmia due to sick sinus syndrome or second or third-degree atrioventricular block;
16. State of depression (HADS score ≥ 11);
17. Other contraindication to any of the study treatments;
18. Inability for the patient to follow the study schedule;
19. Inability for the patient or the healthcare team to perform the treatment within 2 weeks;
20. Pregnant or breastfeeding women, women who are able to conceive and who do not use a highly effective method of contraception during the trial and for at least 1 month after the end of treatment ;
21. Patient under guardianship or curatorship.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Pain assessment using Numerical Pain Scale (END) | 8 weeks after treatment initiation, or the closest measurement within +/- 1 week if the 8-week data is missing.
  The primary outcome measure is pain assessed by self-evaluation using the Numerical Pain Scale (END) ranging from 0 (no pain) to 10 (worst pain imaginable) at rest, evaluated 8 weeks after treatment (or 9 weeks after randomization if treatment was not performed). The patient's self-assessment reflects individual treatment efficacy. In case of treatment interruption due to immediate intolerance or technical issues, the baseline END will be considered for the primary analysis.

SECONDARY OUTCOMES:
Success of Pain Control | Assessed at 8 weeks post-treatment.
  Defined as a reduction in pain of 3 points or more on the Numerical Pain Scale (END) at 8 weeks, with failure indicated in other cases.
Evolution of Pain Scores | Assessed at multiple time points: 1, 2, 4, 6, 8, and 24 weeks.
  Change in pain levels as self-reported by the patient using the END at 1, 2, 4, 6, 8, and 24 weeks after treatment (and at 13, 14, 16, and 18 weeks if treatment is repeated at 12 weeks).
Neuropathic Component Evaluation | Assessed at multiple time points: 1, 2, 4, 6, 8, and 24 weeks.
  Change in neuropathic symptoms assessed via the Neuropathic Pain Symptom Inventory (NPSI) at 1, 2, 4, 6, 8, and 24 weeks after treatment (and at 13, 14, 16, and 18 weeks if treatment is repeated at 12 weeks).
Early Treatment Failure | Assessed at 7 and 14 days post-treatment
  Early failure of local analgesic treatment defined by failure to perform the procedure (due to intolerance or technical issues) or failure to control pain as evaluated at 7 and 14 days post-procedure.
Modification of introduction of New Analgesic Treatment | Assessed at multiple time points: 1, 2, 4, 6, 8, and 24 weeks.
  Documentation of any change in systemic treatement or introduction of new analgesic treatments (e.g., antiepileptics, antidepressants, opioids), with dosages collected at 1, 2, 4, 6, 8, and 24 weeks after treatment (and at 13, 14, 16, and 18 weeks if treatment is repeated).
Adverse Events | From study treatment to 24-weeks follow-up
  Monitoring of adverse events possibly related to the treatment (capsaicin, botulinum toxin type A, or SBP block) during and after the local procedure, graded according to NCI-CTCAE v5.0.
HADS Scale Evaluation | Assessed at baseline, 8 weeks, and 24 weeks.
  Assessment of anxiety and depression using the Hospital Anxiety and Depression Scale (HADS) at baseline, 8 weeks, and 24 weeks.
Quality of Life Assessment | Assessed at baseline, 8 weeks, and 24 weeks.
  Evaluation of health-related quality of life using the SF12 scale at baseline, 8 weeks, and 24 weeks.
Patient General Impression of Change (PGIC) | Assessed at 8 weeks and 24 weeks
  Self-assessment of change in condition from 1 (no change or worse) to 7 (considerable improvement) measured at 8 weeks and 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Didier DELBROUCK, Anesthesiologist, Principal Investigator — Centre Oscar Lambret
Locations (1):
- Centre Oscar Lambret, Lille, Hauts-de-France, France

IPD SHARING:
Plan to Share IPD: No